CLINICAL TRIAL: NCT01370265
Title: Quantification of Myocardial Blood Flow by Positron Emission Tomography and N-13 Ammonia During Regadenoson vs Adenosine Stress
Brief Title: Myocardial Blood Flow by PET and N-13 Ammonia During Regadenoson vs Adenosine Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Principal Investigator, Panithaya Chareonthaitawee, Consultant, Associate Professor, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 10-006377
Record Dates: First submitted 2011-06-06; First posted 2011-06-09 (Estimated); Results first posted 2013-09-05 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Coronary Artery Disease
Keywords: Regadenoson (Lexiscan); PET N-13 ammonia imaging; Myocardial Blood Flow (MBF); Regadenoson Stress
MeSH Terms: conditions — Coronary Artery Disease | interventions — regadenoson; Adenosine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Regadenoson, then Adenosine (Active Comparator): Regadenoson (0.4 mg/5 ml IV) was administered intravenously over 10 seconds, followed immediately by saline flush and N-13 ammonia (10-20 MCi) injection and an additional saline flush in the first intervention period. Adenosine (140 μg/kg/min) was administered intravenously over 6 minutes in the second intervention period (after washout period). Three minutes after the start of adenosine infusion, N-13 ammonia (10-20 mCi) was administered.
  Interventions: Drug: Regadenoson; Drug: Adenosine; Drug: N-13 ammonia
- Adenosine, then Regadenoson (Active Comparator): Adenosine (140 μg/kg/min) was administered intravenously over 6 minutes in the first intervention period. Three minutes after the start of adenosine infusion, N-13 ammonia (10-20 mCi) was administered. After a washout period, Regadenoson (0.4 mg/5 ml IV) was administered intravenously over 10 seconds, followed immediately by saline flush and N-13 ammonia (10-20 MCi) injection and an additional saline flush in the second intervention period.
  Interventions: Drug: Regadenoson; Drug: Adenosine; Drug: N-13 ammonia

INTERVENTIONS:
Drug: Regadenoson — Regadenoson (0.4 mg/5 ml IV) was administered intravenously over 10 seconds, followed immediately by saline flush.
  Other Names: Lexiscan
Drug: Adenosine — Adenosine (140 μg/kg/min) was administered intravenously over 6 minutes.
  Other Names: Adenoscan
Drug: N-13 ammonia — Ammonia N-13 Injection is a radioactive diagnostic agent for Positron Emission Tomography (PET) indicated for diagnostic PET imaging of the myocardium under rest or pharmacologic stress conditions to evaluate myocardial perfusion in patients with suspected or existing coronary artery disease. The N-13 ammonia used in the study was synthesized by the Mayo Cyclotron Facility as per routine institutional clinical protocol.

SUMMARY:
Blockage of the heart arteries (coronary artery disease) can lead to angina (chest pain), heart attacks, heart failure, and/or death. Positron emission tomography (PET) stress myocardial perfusion imaging (MPI) is a powerful tool to help identify blockages in the coronary arteries. During the PET MPI test, a drug is given to mimic the effects of exercise on the heart. The study was done to measure blood flow to the heart using two similar drugs approved to mimic the effects of exercise on the heart in people during a heart stress test. The first drug, called adenosine, has been approved for this use for several decades. The second drug, called regadenoson, was approved in 2008. The investigators were looking at whether the increase in blood flow to the heart with the newer drug (regadenoson) was similar to the increase in blood flow with the older drug (adenosine). This information is important for the use of these drugs in patients and for interpreting the blood flow values.

DETAILED DESCRIPTION:
The hypothesis for this study was that Regadenoson will produce a very similar degree of maximal hyperemia (increased blood flow) as adenosine, the other vasodilator agent. There were only 2 days on study for each subject.

On Day 1 of the study, subjects were interviewed and had a physical exam, including a resting 12-lead electrocardiogram (ECG) to exclude evidence of silent ischemia or myocardial infarction, and other cardiovascular disorders. Subjects were instructed to have a light meal at least 4 hours prior to the PET MPI. Subjects were instructed to abstain from caffeine-containing products for 24 hours prior to the PET scan. Day 1 of the study occurred less than or equal to 4 weeks of Day 2.

On Day 2 of the study, each subject underwent three PET N-13 ammonia (10-20 mCi) dynamic emission acquisitions: resting, regadenoson (0.4 mg/5 mL IV), and adenosine (140 microgram/kg/min; order of regadenoson vs adenosine was randomized according to subject's birth year), and three transmission acquisitions for attenuation correction. Each emission acquisition was separated by 50 min to allow for radioactive decay. At the end of the drug infusions, subjects were monitored for 5-30 min. Based on the known short biological half-lives of these stress agents, the pharmacologic effects of each drug should have dissipated by the time the next drug was administered.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female volunteers over the age of 30.
* Written informed consent will be obtained from each subject.
* Each subject will undergo a history and physical examination

Exclusion Criteria:

* Any cardiovascular or pulmonary symptoms or exam findings
* History of low blood pressure (< 90/50 mmHg)
* Prior cardiac history
* History of hypertension
* History of hyperlipidemia
* History of diabetes mellitus
* History of asthma or chronic obstructive pulmonary disease
* Weight of > 450 pounds
* Chronic kidney disease
* Other serious illness such as cancer
* Current smoking
* Medication use (with the exception of acetaminophen, aspirin, nonsteroidal anti-inflammatory drugs (NSAIDs), and thyroid hormone replacement)
* Illicit drug use
* Prior allergic reaction to adenosine, regadenoson, or aminophylline
* Pregnancy

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-02; Primary Completion 2012-02 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Panithaya Chareonthaitawee, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From June 30 to December 27, 2011 subjects were recruited at Mayo Clinic in Rochester, Minnesota.
Period: Resting Myocardial Blood Flow (MBF)
Arm/Group | Regadenoson, Then Adenosine | Adenosine, Then Regadenoson
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0
Period: Washout Period (50-minute Period Decay)
Arm/Group | Regadenoson, Then Adenosine | Adenosine, Then Regadenoson
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0
Period: First Intervention
Arm/Group | Regadenoson, Then Adenosine | Adenosine, Then Regadenoson
Started | 6 | 6
Completed | 5 | 5
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 1
Period: Washout Period (50-minute Period Decay)
Arm/Group | Regadenoson, Then Adenosine | Adenosine, Then Regadenoson
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Regadenoson, Then Adenosine | Adenosine, Then Regadenoson
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes groups randomized to receive Regadenoson first and Adenosine first.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 12
Age Continuous [Mean (Standard Deviation); unit: years] | 44 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 12
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 26.1 (4.3)

OUTCOME MEASURES:

1. Primary Outcome: Global Hyperemic Myocardial Blood Flow (MBF)
Description: MBF is the rate of blood supplied to the myocardium, or heart muscle. Hyperemic MBF is the rate of myocardial blood flow in the heart muscle during either regadenoson or adenosine stress. Myocardial blood flow was calculated using commercial software (PMOD Technologies, version 2.4).
  The Hyperemic MBF was measured approximately 4 hours after arrival in the PET unit.
Time Frame: Day 2, approximately 4 hours after arrival in positron emission tomography (PET) unit
Population: Analysis per protocol; one participant in each group experienced an ischemic ECG with the first stress drug, and they were withdrawn from the study. This is a per intervention presentation.
Measure: Mean (Standard Deviation); unit: mL/min/gm
Groups:
- Regadenoson: Regadenoson (0.4 mg/5 ml IV) was administered intravenously over 10 seconds, followed immediately by saline flush and N-13 ammonia (10-20 MCi) injection and an additional saline flush.
- Adenosine: Adenosine (140 μg/kg/min) was administered intravenously over 6 minutes. Three minutes after the start of adenosine infusion, N-13 ammonia (10-20 mCi) was administered.
Arm/Group | Regadenoson | Adenosine
Number analyzed (Participants) | 10 | 10
mL/min/gm | 3.1 (1.4) | 3.1 (1.2)
Statistical Analysis 1: Comparison: Regadenoson vs Adenosine; Statistical analysis for hyperemic global MBF between Regadenoson and Adenosine groups (per intervention), alpha level of 0.05; Test type: Superiority or Other; p = 0.14, t-test, 2 sided

2. Secondary Outcome: Resting Global MBF and Resting Segmental MBF
Description: MBF is the rate of blood supplied to the myocardium, or heart muscle. Global Myocardial blood flow was calculated using commercial software (PMOD Technologies, version 2.4).
  Regional MBFs were calculated using commercial software (PMOD Technologies, version 2.4). After the apical and basal slices of the left ventricular myocardium were chosen, the software automatically defined 4 myocardial regions of interest (segments) in the apical planes.
Time Frame: Day 2, approximately 35 minutes after arrival in positron emission tomography (PET) unit
Population: Resting MBF was measured on all subjects prior to the interventions.
Measure: Mean (Standard Deviation); unit: ml/min/gm
Arm/Group | Entire Study Population
Number analyzed (Participants) | 10
ml/min/gm
  Resting Global MBF | 0.8 (0.2)
  Resting Anterior MBF | 0.7 (0.2)
  Resting Septum MBF | 0.9 (0.2)
  Resting Inferior MBF | 0.8 (0.2)
  Resting Lateral MBF | 0.8 (0.2)

3. Secondary Outcome: Global Cardiac Flow Rate
Description: Cardiac Flow Rate was calculated using the equation: hyperemic MBF/resting MBF.
Time Frame: Day 2, approximately 4 hours after arrival in positron emission tomography (PET) unit
Population: Analysis per protocol, one participant in each group experienced an ischemic ECG with the first stress drug, and they were withdrawn from the study. This is a per intervention presentation.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Regadenoson | Adenosine
Number analyzed (Participants) | 10 | 10
ratio | 3.8 (1.5) | 4.0 (1.4)
Statistical Analysis 1: Comparison: Regadenoson vs Adenosine; Statistical analysis for Cardiac Flow Rate (CFR) between Regadenoson and Adenosine groups (per intervention), alpha level of 0.05; Test type: Superiority or Other; p = 0.21, t-test, 2 sided

4. Secondary Outcome: Hyperemic Segmental MBF
Description: Regional MBFs were calculated using commercial software (PMOD Technologies, version 2.4). After the apical and basal slices of the left ventricular myocardium were chosen, the software automatically defined 4 myocardial regions of interest (segments) in the apical planes.
  The hyperemic MBF was measured approximately 4 hours after arrival in the PET unit, depending on the randomization.
Time Frame: Day 2, approximately 4 hours after arrival in positron emission tomography (PET) unit
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL/min/gm
Arm/Group | Regadenoson | Adenosine
Number analyzed (Participants) | 10 | 10
mL/min/gm
  Hyperemic MBF Anterior | 2.5 (0.5) | 2.6 (0.8)
  Hyperemic MBF Septum | 3.1 (0.8) | 3.2 (1.4)
  Hyperemic MBF Inferior | 3.5 (1.6) | 3.6 (1.3)
  Hyperemic MBF Lateral | 2.9 (0.6) | 2.9 (1.1)
Statistical Analysis 1: Comparison: Regadenoson vs Adenosine; Statistical analysis comparing Regadenoson and Adenosine groups (per intervention), for Hyperemic MBF Anterior, alpha level of 0.05; Test type: Superiority or Other; p = 0.57, t-test, 2 sided
Statistical Analysis 2: Comparison: Regadenoson vs Adenosine; Statistical analysis comparing Regadenoson and Adenosine groups (per intervention) for Hyperemic MBF Septum, alpha level of 0.05; Test type: Superiority or Other; p = 0.13, t-test, 2 sided
Statistical Analysis 3: Comparison: Regadenoson vs Adenosine; Statistical analysis comparing Regadenoson and Adenosine groups (per intervention)for Hyperemic MBF Inferior, alpha level of 0.05; Test type: Superiority or Other; p = 0.44, t-test, 2 sided
Statistical Analysis 4: Comparison: Regadenoson vs Adenosine; Statistical analysis comparing Regadenoson and Adenosine groups (per intervention) for Hyperemic MBF Lateral, alpha level of 0.05; Test type: Superiority or Other; p = 0.74, t-test, 2 sided

5. Secondary Outcome: Segmental CFR
Description: CFR was calculated using the equation: hyperemic MBF/resting MBF.
Time Frame: Day 2, approximately 4 hours after arrival in positron emission tomography (PET) unit
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Regadenoson | Adenosine
Number analyzed (Participants) | 10 | 10
ratio
  CFR Anterior | 3.4 (1.1) | 3.7 (1.0)
  CFR Septum | 3.5 (0.7) | 3.6 (1.6)
  CFR Inferior | 4.4 (1.4) | 4.6 (1.3)
  CFR Lateral | 3.9 (1.0) | 4.0 (1.1)
Statistical Analysis 1: Comparison: Regadenoson vs Adenosine; Statistical analysis comparing Regadenoson and Adenosine groups (per intervention for CFR Anterior, alpha level of 0.05; Test type: Superiority or Other; p = 0.78, t-test, 2 sided
Statistical Analysis 2: Comparison: Regadenoson vs Adenosine; Statistical analysis comparing Regadenoson and Adenosine groups (per intervention) for CFR Septum, alpha level of 0.05; Test type: Superiority or Other; p = 0.42, t-test, 2 sided
Statistical Analysis 3: Comparison: Regadenoson vs Adenosine; Statistical analysis comparing Regadenoson and Adenosine groups (per intervention for CFR Inferior, alpha level of 0.05; Test type: Superiority or Other; p = 0.96, t-test, 2 sided
Statistical Analysis 4: Comparison: Regadenoson vs Adenosine; Statistical analysis comparing Regadenoson and Adenosine groups (per intervention) for CFR Lateral, alpha level of 0.05; Test type: Superiority or Other; p = 0.13, t-test, 2 sided

6. Secondary Outcome: Heart Rate (Beats Per Minute (BPM))
Description: The resting heart rate was measured approximately 35 minutes after arrival in the PET unit. The hyperemic heart rate was measured approximately 4 hours after arrival in the PET unit, depending on the randomization.
Time Frame: Day 2, approximately 35 minutes and approximately 4 hours after arrival in the PET unit
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Regadenoson | Adenosine
Number analyzed (Participants) | 10 | 10
bpm
  Resting heart rate | 62 (10) | 60 (9)
  Hyperemic heart rate | 98 (16) | 93 (15)
Statistical Analysis 1: Comparison: Regadenoson vs Adenosine; Statistical analysis comparing Regadenoson and Adenosine groups (per intervention) for resting heart rate, alpha level of 0.05; Test type: Superiority or Other; p = 0.28, t-test, 2 sided
Statistical Analysis 2: Comparison: Regadenoson vs Adenosine; Statistical analysis comparing Regadenoson and Adenosine groups (per intervention) for hyperemic heart rate, alpha level of 0.05; Test type: Superiority or Other; p = 0.51, t-test, 2 sided

7. Secondary Outcome: Hyperemic Blood Pressure (mmHg)
Description: Blood pressure was measured approximately 4 hours after arrival in the PET unit, depending on the randomization.
Time Frame: Day 2, approximately 4 hours after arrival in the PET unit
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Regadenoson | Adenosine
Number analyzed (Participants) | 10 | 10
mmHg
  Systolic | 130 (17) | 132 (23)
  Diastolic | 72 (11) | 75 (17)
Statistical Analysis 1: Comparison: Regadenoson vs Adenosine; Statistical analysis comparing Regadenoson and Adenosine groups (per intervention) for systolic blood pressure, alpha level of 0.05; Test type: Superiority or Other; p = 0.31, t-test, 2 sided
Statistical Analysis 2: Comparison: Regadenoson vs Adenosine; Statistical analysis comparing Regadenoson and Adenosine groups (per intervention) for diastolic blood pressure, alpha level of 0.05; Test type: Superiority or Other; p = 0.08, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Subjects were monitored for adverse events for the time while on study, approximately 4 weeks.
Arm/Group | Regadenoson | Adenosine
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 1/12 | 1/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regadenoson (N=12) | Adenosine (N=12)
Ischemic ECG findings (Cardiac disorders) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
Small sample size; Subjects had no evidence of overt coronary artery disease, occult coronary artery disease affecting stress drug induced hyperemic PET MBF is a possibility; however, hyperemic MBF with both stress drugs would be equally affected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No